CLINICAL TRIAL: NCT04556500
Title: Psychometric Properties of the Turkish Version of the Affordance in the Home Environment for Motor Development-Toddler (AHEMD-T)
Brief Title: Turkish Version of the Affordance in the Home Environment for Motor Development-Toddler (AHEMD-T)
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özge ÇANKAYA, Principal investigator, Hacettepe University
Other Study IDs: GO/12-2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Musculoskeletal Diseases; Genetic Disease; Metabolic Disease; Delays Developmental
MeSH Terms: conditions — Musculoskeletal Diseases; Genetic Diseases, Inborn; Metabolic Diseases; Learning Disabilities

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: investigating the psychometric properties of Turkish Affordance in the Home Environment for Motor Development-Toddler (AHEMD-T) — AHEMD-T will apply to parents who have 18-42 months child/children

SUMMARY:
This study aimed to translate the Affordance in the Home Environment for Motor Development -Toddler (AHEMD-T) into Turkish and examine its psychometric properties.

DETAILED DESCRIPTION:
Child motor development is a complex process which results from the interaction between genetics and the environment. The role of the home as the first environment for child experiences is very important for motor development, especially during infancy. Thus, a more supportive and stimulating environment is associated with more affordances and challenges for infant motor development that may lead to improvement in social and cognitive development.

There is no Turkish questionnaire to evaluate home environment so we aimed to translate the AHEMD-T for using with Turkish children and to investigate psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* Parent who have 18-42 months child
* Volunteers

Exclusion Criteria:

* Parents who are not willing to participate in the study

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Parent who have 18-42 months child
  * Volunteers
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Affordance in the Home Environment for Motor Development-Toddler (AHMED-T) | 6 months
  AHEMD-T consists 67 items with 5 section as outdoor environment, indoor environment, variety of stimulation, gross motor toys and fine motor toys. In addition to simple questions with yes-no responses or a Likert scale, this tool uses descriptive questions and visual examples to guide the respondent in the category of the toys provided. The total score of less than 10 was considered low and a poor assessment of affordance in the home environment. This meant that a few poor-quality opportunities were afforded in the home environment for child motor development. A score of 10-15 was a medium and sufficient assessment with adequate and suitable affordances in the home environment for child motor development. A score of 17-21 was considered high and reflected excellent opportunities in the home environment for child motor development.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Numanoğlu Akbaş, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hwang AW, Liao HF, Granlund M, Simeonsson RJ, Kang LJ, Pan YL. Linkage of ICF-CY codes with environmental factors in studies of developmental outcomes of infants and toddlers with or at risk for motor delays. Disabil Rehabil. 2014;36(2):89-104. doi: 10.3109/09638288.2013.777805. Epub 2013 Apr 17. PMID 23594061
- [Background] Carl G, Priscila M, Cacola. A New Inventory For Assessing Affordance in the Home environment For Motor Development. Early Childhood Edu J 2008;36(1):5-9.